CLINICAL TRIAL: NCT02835885
Title: Parametric Testing of Direct Physiological Effects of Transcutaneous Vagus Nerve Stimulation (tVNS) in Healthy Controls
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Medical University of South Carolina (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: Single
Other Study IDs: Pro00038301
Record Dates: First submitted 2016-07-06; First posted 2016-07-18 (Estimated); Last update posted 2016-07-18 (Estimated); Status verified 2016-06

CONDITIONS: Healthy

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Active tVNS Stimulation (Experimental): Stimulating electrode will be placed on left tragus of subject. Current will be held constant (200% perceptual threshold) while pulse width and frequency are varied.The intervention used to keep current constant is Digitmer High Voltage Stimulator model DS7A TENS unit. Each stimulation period (9 randomized stimulation parameters varying in pulse width and frequency) will last 1 minute with a 3 minute break between each parameter. Physiological data (O2 saturation, blood pressure, breathing rate, and Electrocardiogram (EKG) to measure heart rate ) will be collected continuously.
  Interventions: Device: Digitmer High Voltage Stimulator model DS7A TENS unit
- Sham tVNS Stimulation (Sham Comparator): Stimulating electrode will be placed on left ear lobe of subject for sham tVNS stimulation condition. Current will be held constant (200% perceptual threshold) while pulse width and frequency are varied. The intervention used to keep current constant is Digitmer High Voltage Stimulator model DS7A TENS unit. Each stimulation period (9 randomized stimulation parameters varying in pulse width and frequency) will last 1 minute with a 3 minute break between each parameter. Physiological data (O2 saturation, blood pressure, breathing rate, and Electrocardiogram (EKG) to measure heart rate ) will be collected continuously.
  Interventions: Device: Digitmer High Voltage Stimulator model DS7A TENS unit

INTERVENTIONS:
Device: Digitmer High Voltage Stimulator model DS7A TENS unit

SUMMARY:
The purpose of this study is to determine the feasibility and safety of Transcutaneous Vagus Nerve Stimulation (tVNS) in healthy controls. Tested in healthy subjects (HS) the physiological effects of tVNS at different stimulation parameters. The electrical stimulation variables will be pulse width, frequency, and current. This will be tested in a laboratory setting and will measure tVNS effects on heart rate, respiration rate, blood pressure, and perceived pain. This is a feasibility and small safety study.

Hypothesis: tVNS is feasible and safe

ELIGIBILITY:
Inclusion Criteria:

* Meets none of the Exclusion Criteria

Exclusion Criteria:

* History of seizures, depression, or pain conditions
* Taking any prescription medications (excluding contraceptives and statins)
* History of any ear trauma
* History of heart conditions
* Has a heart pacemaker or artificial valve
* Has a metal implant above the waste
* Is pregnant
* Alcohol Dependence
* Illicit drug use in past 6 months
* History of brain surgery or lesions
* History of loss of consciousness (>15 min)
* Faint at the sight of blood
* Hospitalization or surgeries in past 6 months

Ages: 18 Years to 70 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 15 (Actual)
Dates: Start 2014-11; Primary Completion 2015-08 (Actual)

PRIMARY OUTCOMES:
Change from Baseline Heart Rate Before Each Stimulation Period (1-9) to Post Stimulation Period (1-9) Visit 1 | Total time for Visit 1 (either active or sham condition) is 50 minutes - 9 Stimulation Periods (each 4 minutes long with 90 seconds between)
  There are nine stimulation periods, each with own stimulation parameters that consist of a constant current, pulse width and frequency. Each stimulation period has 1 minute of stimulation (active or sham), followed by 3 minutes of post stimulation baseline recording Each of the stimulation period last 4 minutes with an additional 90 seconds between each Stimulation period. Current will be 200% of the subject's perceptual threshold for each stimulation parameter. The pulse width will be either 100 microseconds (µs), 200 µs, or 500µs. Frequency will be either 1 Hertz (Hz), 10 Hz, or 25 Hz.
  Baseline physiological data,Electrocardiogram (EKG) to measure heart rate in beats/sec will be collected before each stimulation parameter, during stimulation parameter, and post each stimulation parameter.
Change from Baseline Heart Rate Before Each Stimulation Period (1-9) to Post Stimulation Period (1-9) Visit 2 | Total time for Visit 2 (either active or sham condition) is 50 minutes - 9 Stimulation Periods (each 4 minutes long with 90 seconds between)
  There are nine stimulation periods, each with own stimulation parameters that consist of a constant current, pulse width and frequency. Each stimulation period has 1 minute of stimulation (active or sham), followed by 3 minutes of post stimulation baseline recording Each of the stimulation period last 4 minutes with an additional 90 seconds between each Stimulation period. Current will be 200% of the subject's perceptual threshold for each stimulation parameter. The pulse width will be either 100 microseconds (µs), 200 µs, or 500µs. Frequency will be either 1 Hertz (Hz), 10 Hz, or 25 Hz.
  Baseline physiological data,Electrocardiogram (EKG) to measure heart rate in beats/sec will be collected before each stimulation parameter, during stimulation parameter, and post each stimulation parameter.
Change from Baseline O2 Saturation Before Each Stimulation Period (1-9) to Post Stimulation Period (1-9) Visit 1 | Total time for Visit 1 (either active or sham condition) is 50 minutes - 9 Stimulation Periods (each 4 minutes long with 90 seconds between)
  There are nine stimulation periods, each with own stimulation parameters that consist of a constant current, pulse width and frequency. Each stimulation period has 1 minute of stimulation (active or sham), followed by 3 minutes of post stimulation baseline recording Each of the stimulation period last 4 minutes with an additional 90 seconds between each Stimulation period. Current will be 200% of the subject's perceptual threshold for each stimulation parameter. The pulse width will be either 100 microseconds (µs), 200 µs, or 500µs. Frequency will be either 1 Hertz (Hz), 10 Hz, or 25 Hz.
  Baseline physiological data O2 saturation (% oxygen) will be collected before each stimulation parameter, during stimulation parameter, and post each stimulation parameter.
Change from Baseline O2 Saturation Before Each Stimulation Period (1-9) to Post Stimulation Period (1-9) Visit 2 | Total time for Visit 2 (either active or sham condition) is 50 minutes - 9 Stimulation Periods (each 4 minutes long with 90 seconds between)
  There are nine stimulation periods, each with own stimulation parameters that consist of a constant current, pulse width and frequency. Each stimulation period has 1 minute of stimulation (active or sham), followed by 3 minutes of post stimulation baseline recording Each of the stimulation period last 4 minutes with an additional 90 seconds between each Stimulation period. Current will be 200% of the subject's perceptual threshold for each stimulation parameter. The pulse width will be either 100 microseconds (µs), 200 µs, or 500µs. Frequency will be either 1 Hertz (Hz), 10 Hz, or 25 Hz.
  Baseline physiological data O2 saturation (%oxygen) will be collected before each stimulation parameter, during stimulation parameter, and post each stimulation parameter.

SECONDARY OUTCOMES:
Change from Baseline Blood Pressure Before Each Stimulation Period (1-9) to Post Stimulation Period (1-9) Visit 1 | Total time for Visit 1 (either active or sham condition) is 50 minutes - 9 Stimulation Periods (each 4 minutes long with 90 seconds between)
  There are nine stimulation periods, each with own stimulation parameters that consist of a constant current, pulse width and frequency. Each stimulation period has 1 minute of stimulation (active or sham), followed by 3 minutes of post stimulation baseline recording Each of the stimulation period last 4 minutes with an additional 90 seconds between each Stimulation period. Current will be 200% of the subject's perceptual threshold for each stimulation parameter. The pulse width will be either 100 microseconds (µs), 200 µs, or 500µs. Frequency will be either 1 Hertz (Hz), 10 Hz, or 25 Hz.
  Baseline physiological data Blood Pressure (mmHg) will be collected before each stimulation parameter, during stimulation parameter, and post each stimulation parameter.
Change from Baseline Blood Pressure Before Each Stimulation Period (1-9) to Post Stimulation Period (1-9) Visit 2 | Total time for Visit 2 (either active or sham condition) is 50 minutes - 9 Stimulation Periods (each 4 minutes long with 90 seconds between)
  There are nine stimulation periods, each with own stimulation parameters that consist of a constant current, pulse width and frequency. Each stimulation period has 1 minute of stimulation (active or sham), followed by 3 minutes of post stimulation baseline recording Each of the stimulation period last 4 minutes with an additional 90 seconds between each Stimulation period. Current will be 200% of the subject's perceptual threshold for each stimulation parameter. The pulse width will be either 100 microseconds (µs), 200 µs, or 500µs. Frequency will be either 1 Hertz (Hz), 10 Hz, or 25 Hz.
  Baseline physiological data Blood Pressure (mmHg) will be collected before each stimulation parameter, during stimulation parameter, and post each stimulation parameter.
Change from Baseline Breathing Rate Before Each Stimulation Period (1-9) to Post Stimulation Period (1-9) Visit 1 | Total time for Visit 1 (either active or sham condition) is 50 minutes - 9 Stimulation Periods (each 4 minutes long with 90 seconds between)
  There are nine stimulation periods, each with own stimulation parameters that consist of a constant current, pulse width and frequency. Each stimulation period has 1 minute of stimulation (active or sham), followed by 3 minutes of post stimulation baseline recording Each of the stimulation period last 4 minutes with an additional 90 seconds between each Stimulation period. Current will be 200% of the subject's perceptual threshold for each stimulation parameter. The pulse width will be either 100 microseconds (µs), 200 µs, or 500µs. Frequency will be either 1 Hertz (Hz), 10 Hz, or 25 Hz.
  Baseline physiological data breathing rate (%CO2) will be collected before each stimulation parameter, during stimulation parameter, and post each stimulation parameter.
Change from Baseline Breathing Rate Before Each Stimulation Period (1-9) to Post Stimulation Period (1-9) Visit 2 | Total time for Visit 2 (either active or sham condition) is 50 minutes - 9 Stimulation Periods (each 4 minutes long with 90 seconds between)
  There are nine stimulation periods, each with own stimulation parameters that consist of a constant current, pulse width and frequency. Each stimulation period has 1 minute of stimulation (active or sham), followed by 3 minutes of post stimulation baseline recording Each of the stimulation period last 4 minutes with an additional 90 seconds between each Stimulation period. Current will be 200% of the subject's perceptual threshold for each stimulation parameter. The pulse width will be either 100 microseconds (µs), 200 µs, or 500µs. Frequency will be either 1 Hertz (Hz), 10 Hz, or 25 Hz.
  Baseline physiological data breathing rate (%CO2) will be collected before each stimulation parameter, during stimulation parameter, and post each stimulation parameter.

IPD SHARING:
Plan to Share IPD: No